CLINICAL TRIAL: NCT03257748
Title: Effects of Laser Therapy and LED Therapy on Elderly Individuals With Temporomandibular Disorder: a Randomized, Controlled, Double-blind, Clinical Trial
Brief Title: Effects of Laser Therapy and LED Therapy on Elderly Individuals With Temporomandibular Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DTMLU
Record Dates: First submitted 2017-08-11; First posted 2017-08-22 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Laser and LED Therapy on Elderly Individuals With Temporomandibular Disorder
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LED group (Experimental): The groups will be submitted to 12 sessions of phototherapy held twice a week for six weeks, during which only the researcher in charge of programming the phototherapy device will be aware of which treatment is being employed. However, the programmer will not participate in the execution of the treatments, evaluations or data analysis.
  Interventions: Radiation: LED therapy
- Laser group (Experimental): The groups will be submitted to 12 sessions of phototherapy held twice a week for six weeks, during which only the researcher in charge of programming the phototherapy device will be aware of which treatment is being employed. However, the programmer will not participate in the execution of the treatments, evaluations or data analysis.
  Interventions: Radiation: Laser Therapy

INTERVENTIONS:
Radiation: Laser Therapy — The groups will be submitted to 12 sessions of phototherapy held twice a week for six weeks, during which only the researcher in charge of programming the phototherapy device will be aware of which treatment is being employed. However, the programmer will not participate in the execution of the treatments, evaluations or data analysis.
  Arms: Laser group
Radiation: LED therapy — The groups will be submitted to 12 sessions of phototherapy held twice a week for six weeks, during which only the researcher in charge of programming the phototherapy device will be aware of which treatment is being employed. However, the programmer will not participate in the execution of the treatments, evaluations or data analysis.
  Arms: LED group

SUMMARY:
Temporomandibular disorder (TMD) is described as a subgroup of orofacial pain with a set of signs and symptoms that involve the temporomandibular joint, masticatory muscles, ears and neck. TMD can occur unilaterally or bilaterally and approximately 70% of the population is affected with at least one sign. The disorder progresses with orofacial pain, muscle pain involving the masticatory and cervical muscles, joint noises (clicks and pops), joint block, mandibular dysfunction and headache. The etiology can be abnormal occlusion and/or posture, trauma involving local tissues, repetitive microtrauma, parafunctional habits and an increase in emotional stress. Studies have demonstrated that phototherapy is an efficient option for the treatment of TMD, leading to improvements in pain and orofacial function. The aim of the proposed study is to analyze the effects of low-level laser therapy and light-emitting diode (LED) therapy on pain and function in patients with TMD. Methods: A randomized, controlled, double-blind, clinical trial is proposed, which will involve 80 individuals between 40 and 70 years of age allocated to either a laser group or LED group submitted to twelve sessions of phototherapy. The Research Diagnostic Criteria for TMDs will be used to evaluate all participants. Pain will be measured using the visual analog scale. Orofacial function will be measured based on maximum vertical mandibular movement and muscle tension (determined through palpation of the masseter, temporal, frontal, sternocleidomastoid, suboccipital and trapezius muscles). Electromyographic analysis of the masseter and anterior temporal muscles will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of TMD based on the RDC/TMD;
* Age between 40 and 70 years.

Exclusion Criteria:

* Dentofacial anomalies;
* Currently in orthodontic or orthopedic treatment for the jaw;
* Currently undergoing physical therapy;
* Currently undergoing psychological treatment;
* Use of muscle relaxant or anti-inflammatory agent.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-11-20 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Through study completion, an average of 1 year.
  This scale will be used for the assessment of pain and consists of a 10-cm line with 0 (absence of pain) printed at one end and 10 (debilitating pain) printed at the other end. The participants will be asked to mark a place on the line that represents their current pain intensity. The researcher will subsequently use a ruler to register the distance from zero to obtain a numeric representation of the pain level. These procedures will be performed before and immediately after treatment.

OTHER OUTCOMES:
Visual Analog Scale | Through study completion, an average of 1 year.
  This scale will be used for the assessment of pain and consists of a 10-cm line with 0 (absence of pain) printed at one end and 10 (debilitating pain) printed at the other end. The participants will be asked to mark a place on the line that represents their current pain intensity. The researcher will subsequently use a ruler to register the distance from zero to obtain a numeric representation of the pain level. These procedures will be performed before and immediately after treatment.
Maximum vertical mandibular movement | Through study completion, an average of 1 year.
  Maximum vertical mandibular movement: The volunteer will be instructed to open his/her mouth a wide as possible. Maximum vertical mandibular movement will be measured as the distance between the maxillary and mandibular central incisors determined with the aid of digital calipers. The volunteer will then be instructed to exert pressure on the mandibular teeth with the mouth open and move the mandible to the right and left for the determination of excursion (distance between upper and lower mid points). These procedures will be performed before and immediately after treatment.
Muscle tension | Through study completion, an average of 1 year.
  Muscle tension: Palpation will be performed of the masseter, temporal, frontal, sternocleidomastoid, suboccipital and trapezius muscle. The classification proposed by Jensen et al. will be used, with the following scores: 0 = absence of pain; 1 = mild discomfort; 2 = moderate pain; and 3 = severe pain. These procedures will be performed before and immediately after treatment.
Electromyography | Through study completion, an average of 1 year.
  The electrical signals of the right and left masseter and anterior temporal muscles will be captured. The EMG signal will be determined using a four-channel acquisition system (EMG System do Brasil Ltda.) with a sampling frequency of 2 KHz. The signal will be digitized using an analog-to-digital converter with 16 bits of resolution. The EMGLab (EMG System do Brasil Ltda) will be employed as the acquisition system. These procedures will be performed before and immediately after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra K Bussadori, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- UniNove, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Langella LG, Silva PFC, Costa-Santos L, Goncalves MLL, Motta LJ, Deana AM, Fernandes KPS, Mesquita-Ferrari RA, Bussadori SK. Photobiomodulation versus light-emitting diode (LED) therapy in the treatment of temporomandibular disorder: study protocol for a randomized, controlled clinical trial. Trials. 2018 Jan 26;19(1):71. doi: 10.1186/s13063-018-2444-7. PMID 29373998